CLINICAL TRIAL: NCT06209736
Title: A Phase 2 Proof of Concept Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of OMS906 in Patients With C3 Glomerulopathy (C3G) and Idiopathic Immune Complex-Mediated Glomerulonephritis (ICGN)
Brief Title: Safety and Efficacy Study of OMS906 in Patients With C3G and ICGN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS906-C3G-001
Record Dates: First submitted 2024-01-04; First posted 2024-01-17 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: C3 Glomerulopathy; Idiopathic Immune Complex-Mediated Glomerulonephritis
Keywords: C3G; ICGN

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study Drug OMS906 (Experimental): Repeat-dose OMS906 5 mg/kg IV administration at 4-week intervals
  Interventions: Drug: OMS906 study drug

INTERVENTIONS:
Drug: OMS906 study drug — OMS906 study drug dose 5mg/kg IV administration at 4-week internals
  Other Names: OMS906

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of OMS906 in patients with C3 Glomerulopathy (C3G) and Idiopathic Immune Complex-Mediated Glomerulonephritis (ICGN)

DETAILED DESCRIPTION:
This is a multicenter, open-label, uncontrolled, non-comparative, fixed-dose study. The primary objective is to assess safety and tolerability of OMS906 in patients with C3G or idiopathic ICGN, both complement-mediated disorders. Patients will receive 5 mg/kg administered as intravenous (IV) infusions at 4-week intervals. The study will enroll up to approximately 20 patients with C3G or ICGN. Safety will be evaluated in all patients and by disease cohort. Preliminary efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) will be evaluated by disease cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults 18 years and older.
2. Competent to provide informed consent and has completed informed consent procedures.
3. Diagnosis of C3G, including dense deposit disease, or ICGN confirmed by biopsy within 36 months of screening.
4. Two 24-hour UPCR ≥ 0.8 gm/gm with the 2 collections separated by 14 - 28 days.
5. GFR estimated by the CKD-EPI equation ≥ 45 mL/min/1.73 m2.
6. Serum C3 concentration less than the lower limit of laboratory normal during screening.
7. Must be on stable maximally tolerated or allowed dose of ACE inhibitor or ARB for at least 90 days.
8. If receiving a sodium-glucose co-transporter-2 (SGLT-2) inhibitor, must be on a stable dose for at least 90 days.
9. If receiving mycophenolate mofetil, a mineralocorticoid receptor antagonist, or a corticosteroid, must be on stable dose for at least 90 days.
10. Have current vaccination status for Neisseria meningitidis, Streptococcus pneumonia and Haemophilus influenza (where available) and agree to maintain vaccination throughout the study.

    Patients who have not received these vaccinations at the time of screening may be vaccinated at any time prior to 2 weeks before the first study drug administration. Vaccine serotypes will be chosen by the local standard of care and serotype prevalence.
11. Female patients of child-bearing potential must have a negative highly sensitive pregnancy test at screening and prior to each dose of OMS906.
12. Females must use highly effective birth control* to prevent pregnancy during the clinical trial and for 20 weeks (140 days) following their last dose of study drug.
13. Males must use highly effective birth control* with a female partner to prevent pregnancy during the clinical trial and for 20 weeks (140 days) following their last dose of study drug.

Exclusion Criteria:

1. History of major organ transplant or hematopoietic stem cell/marrow transplant.
2. Have known congenital deficiency of any of complement factors C1q, C1r, C1s, C2 or C4.
3. Have rapidly progressing glomerulonephritis defined as a 50% or greater decline in the eGFR within 3 months with renal biopsy findings of glomerular crescent formation seen in at least 50% of glomeruli.
4. Have renal biopsy findings showing interstitial fibrosis/tubular atrophy of more than 50%.
5. Immunodeficiency or treatment with immunosuppressive agents (except mycophenolate mofetil or corticosteroids at the prednisone equivalent of ≤ 7.5 mg/day in patients with C3G only) within 90 days of screening.
6. Treatment with rituximab within 6 months of screening.
7. Resting blood pressure > 140/90 mmHg during screening.
8. History of any active malignancy within 5 years of screening except non-melanoma skin cancers.
9. History of monoclonal gammopathy of unknown significance or any autoimmune disorder.
10. Elevation of liver function tests, defined as total bilirubin > 2 × upper limit of normal (ULN), direct bilirubin > 1.5 × ULN, and elevated transaminases, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 × ULN.
11. History of any severe hypersensitivity reactions to other monoclonal antibodies or excipients included in the OMS906 preparation.
12. Significant active bacterial or viral infection within the 2 weeks prior to screening including Covid-19 infection.
13. Use of any other complement inhibitor within 6 months prior to the screening visit.
14. Have human immunodeficiency virus, hepatitis B, or untreated hepatitis C infection.
15. Pregnant, planning to become pregnant, or nursing female patient.
16. Recent surgery requiring general anesthesia within the 2 weeks prior to screening or expected to have surgery requiring general anesthesia during the treatment period.
17. History of any significant medical, neurologic, or psychiatric disorder that in the opinion of the investigator would make the patient unsuitable for participation in the study.
18. Treatment with any investigational medicinal product or investigational device within 30 days (or within 5 × its half-life in days, whichever is the longer period) prior to screening, or participation in another concurrent clinical trial involving a therapeutic intervention. Participation in observational and/or registry studies is permitted.
19. Unable or unwilling to comply with the requirements of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
To assess OMS906 5mg/kg IV administration at 4-week intervals in patients with C3G and ICGN. | 48 weeks
  Number of participants with Adverse Events following dosing of OMS906.

SECONDARY OUTCOMES:
Change in proteinuria measured by 24-hour urine protein/creatinine ratio (UPCR). | 12, 24, 48 weeks
  Change from baseline in proteinuria measured as 24-hour UPCR at 12, 24, and 48 weeks.
Change in proteinuria measured by 24-hour urine protein excretion (UPE). | 12, 24, and 48 weeks.
  Change from baseline in proteinuria measured as 24-hour UPE at 12, 24, and 48 weeks.
Change in proteinuria measured as 24-hour urine albumin excretion (UAE). | Time Frame: 12, 24, and 48 weeks.
  Change from baseline in proteinuria measured as 24-hour UAE at 12, 24, and 48 weeks.
Change in proteinuria measured as 24-hour urine albumin/creatinine ratio (UACR). | 12, 24, and 48 weeks.
  Change from baseline in proteinuria measured as 24-hour UACR at 12, 24, and 48 weeks.
Incidence of participants with a change from baseline of estimated glomerular filtration rate (eGFR) calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula at 24 and 48 weeks. | 24 and 48 weeks
  Number and % of participants with a change from baseline of estimated glomerular filtration rate (eGFR) calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula at 24 and 48 weeks.
Incidence of participants with a change from baseline serum creatinine concentration at 24 and 48 weeks. | 24 and 48 weeks
  Number and % of participants with a change from baseline serum creatinine concentration at 24 and 48 weeks.
Pharmacodynamics (PD) of multiple-dose administration of OMS906. | 48 weeks
  Mature Complement Factor D (CFD) concentration.
Pharmacokinetics (PK) of multiple-dose administration of OMS906 - Cmax. | 48 weeks
  PK parameters including OMS906 maximum concentration - peak plasma concentration (Cmax).
Pharmacokinetics (PK) of multiple-dose administration of OMS906 - AUC. | 48 weeks
  PK parameters - Area under the plasma concentration vs time curve (AUC).
OMS906 anti-drug antibodies (ADA). | 48 weeks
  Number of patients with measurable ADA.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Whitaker, MD, Study Director — Omeros Corporation
Locations (6):
- Lithuania (2):
  - Omeros Investigational Site, Kaunas
  - Omeros Investigational Site, Vilnius
- Omeros Investigational Site, Auckland, New Zealand
- Omeros Investigational Site, Lodz, Poland
- United Kingdom (2):
  - Omeros Investigational Site, Leicester
  - Omeros Investigational Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No